CLINICAL TRIAL: NCT05358054
Title: Comparison of Mulligan Mobilization With Movement and Progressive Strengthening Exercises in Patients With Lateral Epicondylitis
Brief Title: Mobilization With Movement and Progressive Strengthening Exercises in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00769 Amman Ullah Nazir
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Lateral Epicondylitis
Keywords: Mobilization with movement, PRE, PRTEE, VAS, HD.
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Experimental): GROUP A
  Interventions: Other: Mobilization with movement lateral Glides and Conventional Physiotherapy; Other: Progressive Resistance Exercises and Conventional Physiotherapy
- GROUP B (Experimental): GROUP B
  Interventions: Other: Mobilization with movement lateral Glides and Conventional Physiotherapy; Other: Progressive Resistance Exercises and Conventional Physiotherapy

INTERVENTIONS:
Other: Mobilization with movement lateral Glides and Conventional Physiotherapy — (The Mobilization with movement technique is(lateral glide) applied to the patient by a physiotherapist to patients at supine level position.
  First we identify pain free region each patients. The lateral humerus above the condyle of elbow joint are fixed by therapist. Then therapist ask to patients perform the active movement ten times. The same procedure repeats number of 3 sets, 10 number of repetition. The rest of interval fifteen to twenty seconds with in the sets Grip strength (pain Free Strength ) was evaluated in kilogram using a dynamometer. The measurements using dynamometer patients posture is erect sit position , the elbow at 90 degree flexion , shoulder would be abducted , rest of joint forearm and wrist in neutral during measurements.
  conventional therapy list of conventional physiotherapy are therapeutic ultrasound , deep transverse friction massage and stretching
Other: Progressive Resistance Exercises and Conventional Physiotherapy — 4 STEPS Progressive resistive EXERCISES have a 4 step to application Step 1 Clenching fist strongly, resisted wrist Flexion, Extension, wrist rotation with a stick) Step 2 The therapeutic band exercised performed at wrist Flexion(WF), Wrist Extension(WE), Wrist Ulnar Deviation(WED) , and Wrist Radial Deviation(WRD).Step 3 Patient asked to perform combined wrist rotatory movements using e.g. table top as a support. Step 4 Soft ball compressing exercises, Transferring buttons from cup into another, Twisting a towel into the roll, Hand Rotating both directions at table AND CONVENTIONAL PHYSIOTHERAPY and list of conventional physiotherapy are therapeutic ultrasound , deep transverse friction massage and stretching

SUMMARY:
The purpose of the study is to compare the mobilization with movement and progressive strengthening exercises in individuals with lateral epicondylitis on VAS, PRTEE and Hand Grip strength . A randomized clinical trial was conducted at Bone and Joint center and Khyaban medical center, Rawalpindi. The sample size was 40 calculated through open-epi tool . The participants were divided into two groups each having 20 participants. The study duration was six months. Sampling technique applied was Purposive sampling for recruitment and group randomization using enveloped sealed. Only 20 to 60 years participants with chronic lateral epicondylitis included in that study . Tools used in this study are SELF STRUCTURE QUESTIONNAIRE, VAS visual analogue scale range is 0 TO 10 O is no pain 10 is unbearable pain , PRTEE patient ratted tennis elbow evaluation 15 questionnaire form 3 sub-scale total 100 scores 0 is best 100 is worst, hand held Dynamo-meter , Data was collected before and immediately after the application of interventions. Data analyzed through SPSS version 21.

DETAILED DESCRIPTION:
Epicondylitis is common in persons who frequently overuse the upper arm, particularly with activities that involve rotation of the arm with flexion and extension.

Anyone who performs repetitive movements involving extension of the wrist or hand for at least two hours a day, which can include anyone sitting at a computer and using a mouse. Professional who are commonly effected are Tennis Players, Squash Players, Badminton Players ,Painters, Plumbers, Computer user and Musician.

Lateral Epicondylitis affect the extensor muscle around elbow also common for extensor type pathology.

Evidence suggests that Prevalence of Tennis elbow generally affects about 1 to 3 % general population from 35 to 50 years .

Lateral epicondylitis of young age around 20 years is usually due to overused sustained pressure during laptop working and it mainly effect the dominant hand usually right hand.

The condition tends to affect men and women equally. The annual incidence is one to three percent in the United States. Despite the condition being commonly referred to as tennis elbow, tennis players make up only 10% of the patient population. Half of the tennis players develop pain around the elbow, of which 75% represent true tennis elbow.

Diagnosis of Lateral Epicondylitis is based on the palpation around lateral elbow region , found local tenderness around lateral epicondyle region and Cozen test , Mill,s test.

Literature review: A systematic and evidence based search of relevant literature was performed by utilizing PubMed and Google Scholar as search engines and the key words used were Lateral Epicondylitis , Tennis Elbow, PRE, Strengthening exercises ,VAS, exercises programme for tennis elbow, .The purpose of the literature review is to find out the pre-existing literature regarding the mobilization with movement and PRE interventions for Lateral Epicondylitis .

In 2020, The Effects of Mulligan's Mobilization with movement technique in patients with lateral epicondylitis. MWM is secure and shows efficacy in terms of outcomes at elbow pain (VAS) , Functional Capacity( FC) PRTEE, and Pain less maximized grip strength, these all parameters showed significant improvement.

An experimental study was conducted in 2017 Effects of progressive strengthening exercises in chronic lateral epicondylitis. The group receiving PRE showed significant improvement in study variables (VAS, PRTEE, Grip Strength). The group which performed PRE and conventional physiotherapy showed greater improvement than alone conventional treatment for lateral epicondylitis .

RCT was conducted in 2016 MWM compared to supervised exercises in patients with lateral epicondylitis. This study showed that the group with mulligan technique's showed effectiveness in term of reduction of pain and improved Grip Hand Strength (GHS) as compared with supervised exercise program group.

An Intervention Comparative study was conducted in 2013 Effectiveness of MWM compared with manipulation of wrist in lateral epicondylitis . The variables were pain , Functional disability recorded by VAS, PRTEE, and Hand Dynamo-meter .This study showed that mulligan mobilization plus conventional treatment was much more effective in treatment of tennis elbow .

RCT was conducted in 2012 MWM as adjunct to conventional physiotherapy in treatment of chronic lateral epicondylitis stated that Mobilization with movement group showed significant improvement in pain reduction at VAS and improved Pain Free Grip Strength .

ELIGIBILITY:
Inclusion Criteria:

* During Palpation found local tenderness over lateral side of epicondyle.
* Diagnosed clinically minimum 3 month duration from orthopedic doctors/ department.
* Positive Mills test or Cozen test.

Exclusion Criteria:

* Traumatic injury
* Any Positive history of ligament or tendon tear grade 3
* Any kind of surgery around elbow past two months
* Any History of systemic diseases
* Any kind of neurological conditions like stroke, MS, CVA.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1st Day
  A Visual Analogue Scale is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.The VAS is pain numeric scale to find out pain intensity and pain level perceived by patients. The VAS is a subjective type pain scale measured the acute and chronic level pain. Score are marked between no pain and worst pain ( zero to 10)
Patients Related Tennis Elbow Evaluation | 1st Day
  Measurements the patient functional status its 15 questionnaires In PRTEE First subscale is The Pain Subscale detail is 5 items Maximum or best score is 0 and worst score is 50 The Second Subscale or PRTEE is The Specific Activities detail is 6 items with finest score is 0 and least score is 60 The third one subscale of PRTEE the Usual Activities sub part 4 items with superior score is 0 and least score is 40. Third Fourth Part of PRTEE is The Function Subscale detail is performance bases specific activities and usual or regular activities Add up to specific or regular activities divided by 2 Maximum best score or prime score is 0 and least score is 50 Total detail Score of PRTEE is = Pain Subscale + Function Subscale Best Score= 0 Worst Score = 100 (pain and disability contribute equally to score)
Hand Dynamometer Maximum Grip Strength | 1st day
  A dynamometer with high accuracy and sensitivity has recently been developed to assess grip strength. It provides maximal isometric grip strength measured.Many sports activities hand dynamometer is used to find out athlete performance around hand and forearm muscle strength.
  Sports, like baseball and tennis, where the hand is utilized for tossing or lifting make use of dynamometers to test hand strength

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScPT, Principal Investigator — Riphah International University
Locations (1):
- Bone and joints centre, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwapisz A, Prabhakar S, Compagnoni R, Sibilska A, Randelli P. Platelet-Rich Plasma for Elbow Pathologies: a Descriptive Review of Current Literature. Curr Rev Musculoskelet Med. 2018 Dec;11(4):598-606. doi: 10.1007/s12178-018-9520-1. PMID 30255288
- [Background] Greenberg JA. Endobutton repair of distal biceps tendon ruptures. J Hand Surg Am. 2009 Oct;34(8):1541-8. doi: 10.1016/j.jhsa.2009.05.021. PMID 19801110
- [Background] Coombes BK, Bisset L, Vicenzino B. Management of Lateral Elbow Tendinopathy: One Size Does Not Fit All. J Orthop Sports Phys Ther. 2015 Nov;45(11):938-49. doi: 10.2519/jospt.2015.5841. Epub 2015 Sep 17. PMID 26381484
- [Background] Degen RM, Conti MS, Camp CL, Altchek DW, Dines JS, Werner BC. Epidemiology and Disease Burden of Lateral Epicondylitis in the USA: Analysis of 85,318 Patients. HSS J. 2018 Feb;14(1):9-14. doi: 10.1007/s11420-017-9559-3. Epub 2017 Jun 5. PMID 29398988
- [Background] Reyhan AC, Sindel D, Dereli EE. The effects of Mulligan's mobilization with movement technique in patients with lateral epicondylitis. J Back Musculoskelet Rehabil. 2020;33(1):99-107. doi: 10.3233/BMR-181135. PMID 31104005
- [Background] Upadhyay S, Shukla Y, Patel KK. Effects of progressive strengthening exercises in chronic lateral epicondylitis. Int J Health Sci Res. 2017;7(4):244-57.
- [Background] Rahman H, Chaturvedi PA, Apparao P, Srithulasi PR. Effectiveness of mulligan mobilisation with movement compared to supervised exercise program in subjects with lateral epicondylitis. Int J Physiotherapy Res. 2016;4(2):1394-400.
- [Background] Patel N. Effectiveness of mobilization with movement of elbow compared with manipulation of wrist in patients of lateral epicondylitis. Int J Physiother Res. 2013;1(4):177-82.
- [Background] Anap D, Shende M, Khatri S. Mobilization with movement technique as an adjunct to conventional physiotherapy in treatment of chronic lateral epicondylits-a comparative study. J Nov Physiother. 2012;2(121):2. .
- [Background] Lee JH, Kim TH, Lim KB. Effects of eccentric control exercise for wrist extensor and shoulder stabilization exercise on the pain and functions of tennis elbow. J Phys Ther Sci. 2018 Apr;30(4):590-594. doi: 10.1589/jpts.30.590. Epub 2018 Apr 20. PMID 29706713
- [Background] Kim LJ, Choi H, Moon D. Improvement of pain and functional activities in patients with lateral epicondylitis of the elbow by mobilization with movement: a randomized, placebo-controlled pilot study. Journal of Physical Therapy Science. 2012;24(9):787-90.
- [Background] Basak T, Pal TK, Saha MB, Agarwal S, Das T. Comparative Efficacy of Wrist Manipulation, Progressive Exercises and Both Treatments in Patients with Tennis Elbow. International Journal of Health Sciences and Research. 2018;8(4):87-94.
- [Background] Soonsuwan W, Rangkla S. Comparison between effects of radial extracorporeal shock wave therapy and progressive resistive exercise in treatments of chronic lateral elbow tendinosis. Chulalongkorn Medical Journal. 2017;61(2):193-204.
- [Background] Lucado AM, Dale RB, Vincent J, Day JM. Do joint mobilizations assist in the recovery of lateral elbow tendinopathy? A systematic review and meta-analysis. J Hand Ther. 2019 Apr-Jun;32(2):262-276.e1. doi: 10.1016/j.jht.2018.01.010. Epub 2018 Apr 26. PMID 29705077
- [Background] MacDermid JC. The Patient-Rated Tennis Elbow Evaluation (PRTEE) User Manual. Hamilton, Canada: School of Rehabilitation Science, McMaster University. 2007
- [Background] Cassar M-P. Handbook of clinical massage: Churchill Livingstone; 2004.
- [Background] Cadenas-Sanchez C, Sanchez-Delgado G, Martinez-Tellez B, Mora-Gonzalez J, Lof M, Espana-Romero V, Ruiz JR, Ortega FB. Reliability and Validity of Different Models of TKK Hand Dynamometers. Am J Occup Ther. 2016 Jul-Aug;70(4):7004300010. doi: 10.5014/ajot.2016.019117. PMID 27294996
- [Background] Altan L, Ercan I, Konur S. Reliability and validity of Turkish version of the patient rated tennis elbow evaluation. Rheumatol Int. 2010 Jun;30(8):1049-54. doi: 10.1007/s00296-009-1101-6. Epub 2009 Aug 26. PMID 19707766
- [Background] Thong ISK, Jensen MP, Miro J, Tan G. The validity of pain intensity measures: what do the NRS, VAS, VRS, and FPS-R measure? Scand J Pain. 2018 Jan 26;18(1):99-107. doi: 10.1515/sjpain-2018-0012. PMID 29794282
- [Background] Amro A, Diener I, Isra'M H, Shalabi AI, Dua'I I. The effects of Mulligan mobilisation with movement and taping techniques on pain, grip strength, and function in patients with lateral epicondylitis. Hong Kong Physiotherapy Journal. 2010;28(1):19-23
- [Background] Rees JD, Maffulli N, Cook J. Management of tendinopathy. Am J Sports Med. 2009 Sep;37(9):1855-67. doi: 10.1177/0363546508324283. Epub 2009 Feb 2. PMID 19188560
- [Background] Ahmad Z, Siddiqui N, Malik SS, Abdus-Samee M, Tytherleigh-Strong G, Rushton N. Lateral epicondylitis: a review of pathology and management. Bone Joint J. 2013 Sep;95-B(9):1158-64. doi: 10.1302/0301-620X.95B9.29285. PMID 23997125
- [Background] Kongmalai P, Chanlalit C. Demographic Causes of Chronic Lateral Elbow Pain along Arthroscopic Criteria. J Med Assoc Thai. 2016 Nov;99 Suppl 8:S79-S83. PMID 29901918
- [Background] Fekri L, Rezvani A, Karimi N, Ezzati K. The Effect of Low-Power and High-Power Laser Therapy on Pain, Tenderness and Grip Force of the Patients with Tennis Elbow. Pharma-cophores. 2019;10(3):89-95.
- [Background] )-Padasala M, Sharmila B, Bhatt H, D'Onofrio R. Comparison of efficacy of the eccentric concentric training of wrist extensors with static stretching versus eccentric concentric training with supinator strengthening in patients with tennis elbow: A randomized clinical trial.
- [Background] Uygur E, Aktas B, Ozkut A, Erinc S, Yilmazoglu EG. Dry needling in lateral epicondylitis: a prospective controlled study. Int Orthop. 2017 Nov;41(11):2321-2325. doi: 10.1007/s00264-017-3604-1. Epub 2017 Aug 21. PMID 28828509
- [Background] Shaheen H, Alarab A, Ahmad MS. Effectiveness of therapeutic ultrasound and kinesio tape in treatment of tennis elbow. J Nov Physiother Rehabil. 2019;3:25-33.
- [Background] Abbott JH, Patla CE, Jensen RH. The initial effects of an elbow mobilization with movement technique on grip strength in subjects with lateral epicondylalgia. Man Ther. 2001 Aug;6(3):163-9. doi: 10.1054/math.2001.0408. PMID 11527456
- [Background] Buchbinder R, Green SE, Youd JM, Assendelft WJ, Barnsley L, Smidt N. Shock wave therapy for lateral elbow pain. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD003524. doi: 10.1002/14651858.CD003524.pub2. PMID 16235324
- [Background] Khan MK. Effectiveness of Autologous Blood Injection in Patients with Lateral Epicondylitis (Tennis Elbow). Ophthalmology. 2014;12(2):159.
- [Background] Struijs PA, Smidt N, Arola H, Dijk vC, Buchbinder R, Assendelft WJ. Orthotic devices for the treatment of tennis elbow. Cochrane Database Syst Rev. 2002;(1):CD001821. doi: 10.1002/14651858.CD001821. PMID 11869609